CLINICAL TRIAL: NCT06713538
Title: Impact of a Standardized Equine Mediation Program on the Evolution of the Psycho-behavioral Profile of Adults With Traumatic Brain Injuries Experiencing Impaired Quality of Life.
Brief Title: Impact of a Standardized Equine Mediation Program on the Evolution of the Psycho-behavioral Profile of Adults With Traumatic Brain Injuries Experiencing Impaired Quality of Life (EPONA).
Acronym: EPONA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital La Musse (Other)
Collaborators: Institut Français du Cheval et de l'Equitation IFCE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-A02966-51
Record Dates: First submitted 2024-11-25; First posted 2024-12-03 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Traumatic Brain Injury (TBI) Patients; Equine-assisted Therapy; Cognitive Disorders; Quality of Life
Keywords: Traumatic Brain Injury; Equine Mediation; Cognitive profile; Quality of life
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognitive Dysfunction | interventions — Equine-Assisted Therapy; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): The experimental setup corresponds to a standardized and progressive program of 12 sessions (2 sessions of 90 minutes per week for 6 weeks) of ground work with the horse. These sessions will be protocolized and themed, addressing psycho-behavioral issues commonly found in traumatic brain injury patients (emotion management, strategy development, problem-solving, analysis and interpretation of others' behavior, etc.).
  Interventions: Other: Equine assisted therapy
- Control group (Active Comparator): The control setup is based on global recommendations for physical activity for health (WHO), which advise 150 to 300 minutes of moderate endurance activity per week for a positive impact on physical, cognitive, and psychological health for the 18-65 age group.
  Following these recommendations, the subjects will independently carry out 12 sessions (2 sessions of 90 minutes per week for 6 weeks) of moderate-intensity physical activity. The endurance activity should be performed according to the patient's capabilities and fatigue levels.
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Equine assisted therapy — The intervention will last for 12 sessions, with two 1.5-hour sessions per week. The program is offered to patients in addition to their usual daily schedule. These 12 sessions will be organized as follows:
  Arms: Experimental group
Other: Physical activity — The subjects will independently carry out 12 sessions (2 sessions of 90 minutes per week for 6 weeks) of moderate-intensity physical activity. The endurance activity should be performed according to the patient's capabilities and fatigue levels.
  Arms: Control group

SUMMARY:
In France, 155,000 traumatic brain injuries (TBIs) are treated annually, representing a major public health challenge. The sequelae vary depending on the lesions and include a range of motor disorders as well as complex cognitive and psycho-behavioral impairments that significantly affect autonomy. Psycho-behavioral disorders are present in 75% of cases and hinder the process of social reintegration. The relationships between quality of life, social functioning, and psycho-behavioral profiles raise significant questions within the scientific and medical communities, emphasizing the need for the development of specific care programs for this population.

While non-pharmacological interventions are recommended as a first-line approach at all stages of care, existing therapeutic programs have not demonstrated sufficient effectiveness. As maintaining TBI patients within their communities becomes a priority, aligned with ministerial and HAS (French National Health Authority) recommendations, equine mediation appears to hold significant potential, particularly for addressing psycho-behavioral disorders. These therapeutic techniques have gained considerable traction in recent years, with literature reviews indicating effectiveness across diverse populations (e.g., Autism, Mental Health). However, to our knowledge, no studies have evaluated the potential benefits of equine mediation for TBI patients.

In light of these observations, the EPONA study aims to assess the impact of a standardized horse-assisted therapeutic program on the evolution of the psycho-behavioral profile of TBI patients. The secondary objectives of the study are to measure the impact of this program on the evolution of motor and cognitive profiles, psychological pain, the level of autonomy, social participation, and quality of life.

The primary judgment criterion evaluates the psycho-behavioral profile Brief-A Behavioral Regulation Index Roth 2005 The secondary judgment criteria evaluate impairments activity limitations and participation restrictions For impairments we analyze the cognitive profile with the questionnaire Brief-A Roth 2005 the balance via the Timed Up and Go test the psychological pain with the Rosenberg Self-Esteem Scale Rosenberg 1965 and anxiety via the Hospital Anxiety and Depression Scale Zigmond 1983 For activity limitations we evaluate walking with the Six-Minute Walk Test Guyatt 1985 as well as the level of functional independence Calmels 2009 For participation restrictions we evaluate social participation with the MHAVIE scale Fougeyrollas 2003 as well as quality of life using the QoLIBRI Von Steinbüchel 2005 and CSQ-8 Larsen 1979 scales.

For this single-blind randomized study, 50 traumatic brain injury subjects will be recruited at the Hôpital de la Musse Saint Sébastien de Morsent. Depending on the randomization, patients will be assigned either to the experimental group or the control group. For the experimental group, patients will undergo 12 sessions of equine mediation, with 2 sessions of 90 minutes per week for 6 weeks. For the control group, patients will undergo 12 sessions of physical activity, with 2 sessions of 90 minutes per week for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years.
* Presenting a traumatic brain injury with a non-progressive lesion that occurred at least three months ago (identified using the Neurobehavioural Rating Scale Revised (NRS-R))
* Patients with mild to severe psycho-behavioral disorders
* Subjects must be autonomous for mobility (with or without technical assistance)
* Must not be allergic to horses.
* Able to remain in a seated and standing position (with or without technical assistance).
* Have at least one functional upper limb (to interact with the horse).
* A cognitive level equivalent to primary school (CM1/CM2) enabling the completion of questionnaires.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Individuals in emergency situations
* Individuals participating simultaneously in another study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of psycho-behavioral profile | Pre-test (before intervention), Post-test (immediately after intervention) and Post-test 2 (3months after intervention)
  The psycho-behavioral profile of the patient will be assessed using the Behavior Rating Inventory of Executive Function-Adult Version (Brief-A).

SECONDARY OUTCOMES:
Evaluation of balance | Pre-test (before intervention), Post-test (immediately after intervention) and Post-test 2 (3months after intervention)
  Evaluation of balance using the Timed Up and Go (TUG) test, which assesses the static and dynamic balance of patients and helps predict their risk of falling.
Evaluation of Self-Esteem - Rosenberg | Pre-test (before intervention), Post-test (immediately after intervention) and Post-test 2 (3months after intervention)
  Evaluation of Self-Esteem is carried out using the Rosenberg Scale. The score on this scale ranges from 10 to 40. The lower the score, the lower the self-esteem.
Evaluation of Anxiety and depression | Pre-test (before intervention), Post-test (immediately after intervention) and Post-test2 (3months after intervention)
  Evaluation of Anxiety and depression is carried out using the Hospital Anxiety and Depression Scale (HADS). Seven questions relate to anxiety (total A) and seven to depression (total D), giving two scores (maximum score for each = 21). The higher the scores, the more anxious and depressed the patient.
Evaluation of gait | Pre-test (before intervention), Post-test (immediately after intervention) and Post-test 2 (3months after intervention)
  The patients' walking ability is evaluated using the 6-Minute Walk Test.
Evaluation of functional independence | Pre-test (before intervention), Post-test (immediately after intervention) and Post-test 2 (3months after intervention)
  Evaluation of functional independence is assessed using the Functional Independence Measure (FIM).
Evaluation of social participation | Pre-test (before intervention), Post-test (immediately after intervention) and Post-test 2 (3months after intervention)
  Evaluation of social participation is typically assessed using the measuring lifestyle habits (MHAVIE) scale. Each item is scored from 0 to 9, with a score of zero indicating total disability or interruption of participation, and a score of nine indicating optimal participation. The total LIFE-HM score is obtained by adding up the scores for each item, then dividing by the number of items (calculating an average). The higher the score, the greater the patient's optimal level of participation.
Evaluation of quality of life | Pre-test (before intervention), Post-test (immediately after intervention) and Post-test 2 (3months after intervention)
  Evaluation of quality of life is typically assessed using the Quality of Life in Brain Injury (QoLIBRI) scale, which is designed specifically for individuals with brain injuries. The QOLIBRI questionnaire comprises 37 items rated from 1 to 5. The total score is divided by the number of items to calculate the average. The higher the average, the worse the patient's quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital La Musse, Saint-Sébastien-de-Morsent, France

IPD SHARING:
Plan to Share IPD: Undecided